CLINICAL TRIAL: NCT00709592
Title: Reduced Intensity Myeloablative Total Body Irradiation and Thymoglobulin Followed by Allogeneic Peripheral Blood Stem Cell Transplantation
Brief Title: Reduced Intensity Total Body Irradiation + Thymoglobulin Followed by Allogeneic PBSCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-11561; NCI-2011-01698 (Other: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Results first posted 2015-02-12 (Estimated); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Non-Hodgkin's Lymphoma; Leukemia; Multiple Myeloma; Acute Myeloid Leukemia; Hodgkin Lymphoma; Chronic Lymphocytic Leukemia; Chronic Myelogenous Leukemia; Myelodysplastic Syndrome
Keywords: total body irradiation; Allogeneic Peripheral Blood Stem Cell Transplantation; thymoglobulin
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia; Multiple Myeloma; Leukemia, Myeloid, Acute; Hodgkin Disease; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myelodysplastic Syndromes | interventions — thymoglobulin; Antilymphocyte Serum; Whole-Body Irradiation; Peripheral Blood Stem Cell Transplantation; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ATG 1.7 mg/kg, TBI, transplant (Experimental): (Rabbit-ATG;Thymoglobulin,Genzyme) ATG 5.1 mg/kg in three divided doses (1.7 mg/kg/d) given over three days (day -9 to -7) followed by 450 cGy TBI and tacrolimus plus MMF GVHD prophylaxis. Patients receive lower dose anti-thymocyte globulin IV on days -9 to -7. Patients undergo total-body radiation (TBI) twice daily (BID) on day -1 and once daily (QD) on day 0. Patients then undergo peripheral blood stem cells or bone marrow transplant on day 0. GRAFT-VERSUS-HOST DISEASE PROPHYLAXIS: patients receive tacrolimus orally (PO) on days -2 to 90-120 with taper for 2 months, and mycophenolate mofetil (MMF) PO BID on days 0-30.
  Interventions: Biological: Thymoglobulin; Radiation: Total-Body Irradiation; Procedure: Allogeneic PBSCT or BMT; Drug: Tacrolimus; Drug: Mycophenolate Mofetil
- ATG 2.5 mg/kg/d, TBI, transplant (Experimental): (Rabbit-ATG;Thymoglobulin,Genzyme) ATG 7.5 mg/kg in three divided doses (2.5 mg/kg/d) given over three days (day -9 to -7) followed by 450 cGy TBI and tacrolimus plus MMF GVHD prophylaxis. Patients receive higher dose anti-thymocyte globulin intravenously (IV) on days -9 to -7. Patients undergo total-body radiation (TBI) twice daily (BID) on day -1 and once daily (QD) on day 0. Patients then undergo peripheral blood stem cells or bone marrow transplant on day 0. GRAFT-VERSUS-HOST DISEASE PROPHYLAXIS: patients receive tacrolimus orally (PO) on days -2 to 90-120 with taper for 2 months, and mycophenolate mofetil (MMF) PO BID on days 0-30.
  Interventions: Biological: Thymoglobulin; Radiation: Total-Body Irradiation; Procedure: Allogeneic PBSCT or BMT; Drug: Tacrolimus; Drug: Mycophenolate Mofetil

INTERVENTIONS:
Biological: Thymoglobulin — Patients eligible for participation in this study will be randomized between receiving rabbit ATG for 3 days. Thymoglobulin will be administered according to VCU BMT standard of care starting day -9 and continued daily through day -7.
  Other Names: anti-thymocyte globulin (rabbit); ATG; Genzyme; anti-thymocyte globulin; Rabbit; Rabbit-ATG
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: Whole-Body Irradiation; Total Body Irradiation [TBI]
Procedure: Allogeneic PBSCT or BMT — Undergo allogeneic PBSCT or BMT
  Other Names: PBPC transplantation; Peripheral Blood Progenitor Cell Transplantation; Peripheral Blood Stem Cell Transplantation [Allogenic PBSCT]; Allogeneic Bone Marrow Transplantation [BMT]; Allogeneic BMT; Allogeneic Hematopoietic Stem Cell Transplantation; HSCT
Drug: Tacrolimus — Given PO
  Other Names: Fujimycin; Hecoria; Prograf; Protopic
Drug: Mycophenolate Mofetil — Given PO
  Other Names: CellCept; MMF

SUMMARY:
One of two different doses of thymoglobulin will allow bone marrow engraftment with minimal Graft-versus-Host Disease and allow adequate immune response to allow the transplanted stem cells to replace the tumor cells.

DETAILED DESCRIPTION:
This randomized phase II trial studies how well giving low dose total-body irradiation (TBI) with anti-thymocyte globulin followed by donor peripheral blood stem cell transplant (PBSCT) works in treating patients with hematologic malignancies. Giving reduced intensity total-body irradiation and anti-thymocyte globulin before a donor peripheral blood stem cell transplant helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving total-body irradiation together with antithymocyte globulin before transplant may stop this from happening.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hematological malignancies for which allogeneic stem cell transplantation indicated including non-Hodgkin lymphoma (NHL), multiple myeloma (MM), acute myeloid leukemia (AML), Hodgkin lymphoma (HD), chronic lymphocytic leukemia (CLL), chronic myelogenous leukemia (CML), and myelodysplastic syndrome (MDS)
* Patients with HLA compatible related or unrelated stem cell donor, willing and able to serve as an allogenic HSC donor. Unrelated donors have to be matched at HLA-A, B, C and DRB1 loci. A single locus mismatch will be tolerated in the event a more closely matched donor is not available.
* Patients age >/=40 to </=70 with an ECOG performance status < 2
* Patients between 18 and 40 years of age will be eligible only if they have co-morbidities precluding conventional allogeneic transplantation with full intensity myeloablative conditioning
* Adequate cardiac, pulmonary, renal and hepatic function for transplant
* Negative serology for HIV
* Negative serum pregnancy test
* Patients who have received therapeutic radiation to a localized field will be eligible, provided critical structure tolerance doses have not been exceeded
* Patients who have had prior myeloablative autologous transplant will be eligible

Exclusion Criteria:

* Evidence of uncontrolled viral, fungal, bacterial infection
* Evidence of active meningeal or CNS disease
* Prior therapy with rabbit ATG, prior treatment with equine ATG is allowed if more than 3 months ago
* Breast feeding mothers are excluded

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2008-07-21 (Actual); Primary Completion 2014-02-15 (Actual); Study Completion 2017-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amir Toor, MD, Principal Investigator — Massey Cancer Center
Locations (1):
- Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia, United States

REFERENCES:
- See also: VCU Massey Cancer Center — http://www.massey.vcu.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Consecutive patients enrolled have recurrent or high-risk hematologic malignancy, adequate end-organ function and performance status. Patient required to have 7/8 or 8/8 mismatched related donor (MRD) or unrelated donor (URD), with high-resolution typing performed for HLA-A, -B, -C, and -DRB1.
Pre-assignment Details: Randomized to rabbit ATG (Thymoglobulin; Genzyme, Cambridge, MA), 2.5 or 1.7 mg/kg adjusted ideal body weight/day, followed by TBI to a total dose of 4.5 Gy. Methylprednisolone 2 mg/kg given pre-medication for ATG. GVHD prophylaxis was tacrolimus starting at approximately 12 weeks post transplantation.
Groups:
- A:Thymoglobulin: 1.7 mg/kg/Day: 1.7 mg/kg/d thymoglobulin IV d-9 to -7
- B:Thymoglobulin: 2.5 mg/kg/Day: 2.5 mg/kg/d thymoglobulin IV d-9 to d-7
Period: Overall Study
Arm/Group | A:Thymoglobulin: 1.7 mg/kg/Day | B:Thymoglobulin: 2.5 mg/kg/Day
Started | 19 | 23
Completed | 19 | 22
Not Completed | 0 | 1
Not completed — Unable to proceed to transplant | 0 | 1

BASELINE CHARACTERISTICS:
Population: Subjects able to proceed to transplant.
Groups:
- Total: Total of all reporting groups
Arm/Group | A:Thymoglobulin: 1.7 mg/kg/Day | B:Thymoglobulin: 2.5 mg/kg/Day | Total
Number analyzed (Participants) | 19 | 23 | 42
Age, Continuous [Median (Full Range); unit: years] | 57 [44 to 69] | 57 [40 to 68] | 57 [40 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 12 | 15 | 27
Region of Enrollment [Number; unit: participants]
  United States | 19 | 23 | 42

OUTCOME MEASURES:

1. Primary Outcome: The Comparison of Functional Immune Reconstitution at 6-9 Months Following Transplant as Measured by Antibody Response to Vaccination With Inactivated Hepatitis A or B Vaccine.
Description: A positive test result will indicate immune reconstitution, while a negative test results will indicate lack of immune reconstitution. Participants not done (ND) will be counted with the negative (Neg).
Time Frame: Up to 9 months following transplant
Measure: Number; unit: participants
Arm/Group | A:Thymoglobulin: 1.7 mg/kg/Day | B:Thymoglobulin: 2.5 mg/kg/Day
Number analyzed (Participants) | 19 | 22
participants
  Positive | 8 | 3
  Negative/Not Done | 11 | 19

2. Secondary Outcome: Engraftment of Donor Hematopoietic Stem Cells, as Measured by Time in Days to Neutrophil and Platelet Count Recovery Following Allogeneic PBSCT.
Time Frame: Up to 52 weeks post transplant.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | A:Thymoglobulin: 1.7 mg/kg/Day | B:Thymoglobulin: 2.5 mg/kg/Day
Number analyzed (Participants) | 19 | 22
Days | 12 [10 to 37] | 12 [10 to 37]

3. Secondary Outcome: Survival
Time Frame: 2-year survival rate (%)
Measure: Number; unit: percentage of patient surviving
Arm/Group | A:Thymoglobulin: 1.7 mg/kg/Day | B:Thymoglobulin: 2.5 mg/kg/Day
Number analyzed (Participants) | 19 | 22
percentage of patient surviving | 71.3 | 62.4

4. Secondary Outcome: Treatment Related Mortality
Time Frame: Day 100
Measure: Number; unit: percentage of patients
Arm/Group | A:Thymoglobulin: 1.7 mg/kg/Day | B:Thymoglobulin: 2.5 mg/kg/Day
Number analyzed (Participants) | 19 | 22
percentage of patients | 0 | 0

5. Secondary Outcome: Event-free Survival
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Arm/Group | A:Thymoglobulin: 1.7 mg/kg/Day | B:Thymoglobulin: 2.5 mg/kg/Day
Number analyzed (Participants) | 19 | 22
percentage of participants | 62.2 | 44.5

6. Secondary Outcome: Relapse
Description: Patients with different disease relapses was determined according to current clinical standards based on the disease. For example, AML or MDS relapse is determined by a bone marrow biopsy. Multiple myeloma relapse requires a number of labs and/or biopsy to diagnose such as SPEP, UPEP, immunofixation, serum and urine light chains. In lymphoma disease is followed using CT and/or PET scans.
Time Frame: 2 year relapse rate (%)
Measure: Number; unit: Percent patients relapsing
Arm/Group | A:Thymoglobulin: 1.7 mg/kg/Day | B:Thymoglobulin: 2.5 mg/kg/Day
Number analyzed (Participants) | 19 | 22
Percent patients relapsing | 28 | 50

7. Secondary Outcome: Donor Lymphocyte Infusion
Time Frame: 2 year rate of DLI
Measure: Number; unit: percentage of participants
Arm/Group | A:Thymoglobulin: 1.7 mg/kg/Day | B:Thymoglobulin: 2.5 mg/kg/Day
Number analyzed (Participants) | 19 | 22
percentage of participants | 8.9 | 45.5

8. Secondary Outcome: Acute Graft-Versus-Host Disease (GVHD)
Time Frame: 2 year rate (%)
Measure: Number; unit: percentage of participant
Arm/Group | A:Thymoglobulin: 1.7 mg/kg/Day | B:Thymoglobulin: 2.5 mg/kg/Day
Number analyzed (Participants) | 19 | 22
percentage of participant | 27.2 | 4.5

9. Secondary Outcome: Chronic Graft-Versus-Host Disease (GVHD)
Time Frame: 2 year GVHD rate
Measure: Number; unit: percentage of participants
Arm/Group | A:Thymoglobulin: 1.7 mg/kg/Day | B:Thymoglobulin: 2.5 mg/kg/Day
Number analyzed (Participants) | 19 | 22
percentage of participants | 23.8 | 31.8

ADVERSE EVENTS:
Time Frame: All events collected from first patient accrual up to day 180 or relapse for each subject on each arm.
Description: Still collecting SAEs, subjects on trial until death.
Arm/Group | A:Thymoglobulin: 1.7 mg/kg/Day | B:Thymoglobulin: 2.5 mg/kg/Day
Serious Adverse Events (participants affected / at risk) | 7/19 | 12/22
Other Adverse Events (participants affected / at risk) | 19/19 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A:Thymoglobulin: 1.7 mg/kg/Day (N=19) | B:Thymoglobulin: 2.5 mg/kg/Day (N=22)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) — brain
Hepatic (Gastrointestinal disorders) | 2 (2) | 0 (0) — liver
CNS toxicity (Nervous system disorders) | 1 (1) | 1 (1) — brain
Cardiac dysrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Hemorrhagic cystitis (Renal and urinary disorders) | 1 (1) | 1 (1)
Fever with out bacteremia (Infections and infestations) | 2 (2) | 2 (2)
Fever with Bacteremia +/- abscess (Infections and infestations) | 3 (3) | 6 (6)
Intra-abdominal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Brain abscess (Nervous system disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) — vomiting
Renal (Renal and urinary disorders) | 2 (2) | 0 (0)
Hyponatremia (Renal and urinary disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A:Thymoglobulin: 1.7 mg/kg/Day (N=19) | B:Thymoglobulin: 2.5 mg/kg/Day (N=22)
Grade 3 neutropenia (Blood and lymphatic system disorders) | 19 (19) | 22 (22)
Lymphopenia post conditioning (Blood and lymphatic system disorders) | 19 (19) | 22 (22)
Thrombocytopenia (Blood and lymphatic system disorders) | 19 (19) | 22 (22)
Ocular (Eye disorders) | 0 (0) | 2 (2)
Post transplant neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Bacteremia/Fever (Infections and infestations) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0) — UTI

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes